CLINICAL TRIAL: NCT01405378
Title: Combining Transcranial Direct Current Stimulation (tDCS) With Robot Therapy for the Impaired Upper Limb in Stroke Rehabilitation.
Brief Title: Non-invasive Brain Stimulation for People With Stroke
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: University College, London (Other)
Responsible Party: Principal Investigator, Jane Burridge, PhD, Professor, University of Southampton
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Wessex Innovative Grant P09
Record Dates: First submitted 2011-07-21; First posted 2011-07-29 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Robot Therapy and Real Transcranial Direct Current Stimulation (Experimental): This group will involve carrying out robot therapy and real transcranial Direct Current Stimulation (tDCS).
  Interventions: Device: Robot therapy and transcranial direct current stimulation
- Robot Therapy and sham tDCS (Placebo Comparator): Participants will be randomised to group 2 whereby they will carry out the same robot therapy programme however, receiving sham stimulation.
  Interventions: Device: Robot therapy and transcranial direct current stimulation

INTERVENTIONS:
Device: Robot therapy and transcranial direct current stimulation — Administration of Robot Therapy:
  Therapy will be administered by making use of the Armeo Robot. Sessions will involve high-intensity, repetitive, task-oriented movements directed by video screens. Administration of tDCS:
  Anodal tDCS will be administered using a CE marked transcranial Direct Current Stimulator (Newronika Italy). Direct current will be transferred by a saline-soaked pair of surface sponge electrodes (35 cm2).

SUMMARY:
Every five minutes someone in the UK has a stroke. It is the main cause of long-term disability among adults in the UK despite a fall in age-specific stroke incidence, with a growing number of survivors remaining dependent for activities of daily living. While most people with stroke regain walking ability, upper limb problems with no voluntary arm and hand activity, affecting a third of people after stroke, has a poor prognosis. Transcranial direct current stimulation (tDCS) is a non-invasive procedure used to polarise brain regions through the application of weak direct currents and has the potential to develop into a useful aid to treatment strategies in neurorehabilitation. Recent literature into the application of tDCS in people with arm and hand impairments after stroke has shown promising results on upper limb function measures like the Jebsen-Taylor hand function test. Furthermore, a recent pilot study evaluated a six-week training programme combining tDCS with robot-assisted hand training and reported significant improvements in upper limb function. However, the robot in the latter study focused on single-plane distal movements only and long-term effects of the tDCS were not assessed. Recent robotic developments included robots with three rotational degrees-of-freedom for the upper limb, but the effectiveness of this type of robot combined with tDCS in early stroke settings is unknown. Ethical Approval was sought from NHS NRES Committee South Central- Southampton B (Ref: 11/SC/0345) to conduct this study.

ELIGIBILITY:
Inclusion Criteria:

1. Have a confirmed clinical diagnosis of a haemorrhagic or an ischaemic stroke confirmed clinically or by CT, PET or MRI Scan
2. Experienced a single (first) stroke or multiple strokes
3. In the acute, sub-acute or chronic phase of their recovery (the first three to seven days are referred to as the acute phase. The first two weeks to six months are defined as the sub-acute phase, and the chronic phase begins after three or six months (Teismann et al. 2011, Duncan et al. 2003a)
4. Have had a subcortical or cortical stroke
5. Be over the age of 18 years
6. Have any level of upper limb impairment

Exclusion Criteria:

1. A history of epilepsy (TMS studies) due to the fact that TMS could cause an epileptic fit
2. Impaired gross cognitive function; score of less than 24 of the Mini-Mental State Examination (Folstein et al. 1975)
3. Any metal implants in the head including cochlear implants
4. Any another neurological condition apart from stroke
5. Are currently participants in another intervention study using TMS/tDCS

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-10; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Report change in upper limb function from baseline to 8 weeks and 3 months after treatment | Will be used, exactly before commencing training programme (day 1), at the end of the 8 week training programme and at 3 months follow-up
  Measures sensorimotor function of the upper limb (Sanford et al. 1993; Fugl-Meyer et al. 1975)

SECONDARY OUTCOMES:
Report change in cortical excitability from baseline to 8 weeks and 3 months after treatment | Will be used, exactly before commencing training programme (day 1), at the end of the 8 week training programme and at 3 months follow-up
  Corticospinal excitability will be measured by the administration of focal TMS using a figure-of-eight coil to the M1 area of the affected hemisphere. The 'hot spot' will be established by using neuronavigation equipment called Brain Sight (Rogue Research Inc.). The amplitude of the MEPs and recruitment curve of the anterior deltoid (proximal muscle) and extensor digitorum communis (distal muscle) will be subsequently recorded using electromyography.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, University of Southampton, Southampton, United Kingdom